CLINICAL TRIAL: NCT01679717
Title: Postoperative Therapy After Interposition Arthroplasty in CMC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Norwegian Women´s Public Health Association (Other)
Responsible Party: Principal Investigator, Tove Nilsen, Occupational therapist MSc, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H4/2012
Record Dates: First submitted 2012-08-23; First posted 2012-09-06 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Thumb Osteoarthritis
Keywords: Osteoarthritis; CMC1-joint; Postoperative therapy; Interposition arthroplasty of the thumb; Occupational therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early mobilisation after CMC1-surgery (Active Comparator): Mobilisation at two weeks after operation. The participants will wear a soft splint for six weeks.
  Interventions: Other: Early mobilisation after CMC1-surgery
- Conservative treatment after CMC1-surgery (Other): Current standard procedure: Mobilisation at six weeks after operation. The participants will wear a rigid splint for six weeks.
  Interventions: Other: Early mobilisation after CMC1-surgery

INTERVENTIONS:
Other: Early mobilisation after CMC1-surgery — Comparison of early (two weeks) and conservative (six weeks) mobilisation after operation. Comparison of rigid and soft thumb splint.

SUMMARY:
In this randomized controlled trial the investigators want to investigate whether early versus late mobilisation after surgery in the first carpometacarpal joint (CMC1) leads to a faster recovery of hand function. The investigators also want to explore patients' satisfaction with the two different treatment regimes. The participants in the control group will receive the standard treatment at Diakonhjemmet hospital: immobilisation of the thumb in a splint for six weeks. The participants in the intervention group will use a soft splint for six weeks, but will be instructed to remove the splint daily to perform exercises for the thumb. A total of 70 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis in CMC1 diagnosed by radiography and a surgeon.
* Planned surgery(interposition arthroplasty) in CMC1
* Ability to communicate in Norwegian

Exclusion Criteria:

* Surgery involving other joints of the hand in addition to CMC1.
* Previous surgery of the same thumb.
* Other diseases og injuries that could influence hand function.
* Mental or cognitive deficit.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in The Canadian Occupational Performance Measure (COPM) at 3, 6 and 12 months. | Baseline, 3, 6 and 12 months
  The COPM-assessment starts with an interview, addressing patient specific Hand Osteoarthritis (HOA)-related activity limitations within the areas self-care, productivity and leisure. The patient will thereafter rate the five most important activities for performance and satisfaction with performance, on 1 to 10-point scales (higher scores reflect better performance or higher satisfaction). The Norwegian version of the COPM has been tested for validity, reliability and responsiveness and has demonstrated good ability to detect functional changes in HOA.
Change from baseline in Patient satisfaction with the rehabilitation regimen at 3, 6 and 12 months. | Baseline, 3, 6 and 12 months
  Each patient will be asked to complete a Numeric Rating Scale in order to give an opinion about their postoperative treatment regimen (splint-use, hand function, pain in the thumb, thumb movement and satisfaction with the operation).

SECONDARY OUTCOMES:
Measure for activity performance (MAP-hand). | Baseline, 3, 6 and 12 months
  MAP-hand is a questionnaire consisting of questions about 18 standardised activities. The patients will be instructed to score their ability to perform the activities on a scale from 1(No difficulty)to 4 (Not able to do). The Norwegian version of the MAP-hand has been tested for validity, reliability and responsiveness.
Grip force and pinch grip | Baseline, 3, 6 and 12 months
  The electronical instrument Grippit will be used to measure grip force and pinch grip. In Grippit, force recordings in Newtons (N) are displayed on the electronic unit every 0.5 seconds over a period of 10 seconds. The peak and average of the 20 registrations, as well as the final value (last recording) will be recorded.
Joint mobility | Baseline, 3, 6 and 12 months
  * The flexion deficit of fingers 2 - 5 will be assessed by measuring the distance between the distal nail and the proximal crease inside the hand in millimeters.
  * Range of motion in the thumbs metacarpophalangeal and interphalangeal joints will be measured with a goniometer.
  * The palmar abduction of the CMC1 and of the entire thumb will be measured with the Pollexograph.
Pain | Baseline, 3, 6, and 12 months
  Pain will be measured on a numeric rating scale (NRS), (0-10, 0=no pain), by asking the patients to mark the level of pain experienced both while they are resting and during resisted motion when measuring grip force and pinch grip.

OTHER OUTCOMES:
Training diary | Intervention group: 2-6 weeks and 3-4 months. Control group: 6-10 weeks and 3-4 months.
  The patients will be asked to report which date they performed exercises, which exercises they performed and how much pain they experienced after performing the exercises. They will also be encouraged to write down their own comments /reflections regarding the training.

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild Kjeken, Ph.d, Study Chair — Department of Rheumatology, Diakonhjemmet hospital
Locations (1):
- Diakonhjemmet hospital, Oslo, Norway